CLINICAL TRIAL: NCT01974674
Title: Allogeneic Islet Transplantation for the Treatment of Type 1 Diabetes
Acronym: GRIIF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P030415
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Patients With Type 1 Diabetes
Keywords: diabetes; transplantation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic transplantation of intrahepatic islet (Experimental): Allogeneic transplantation of intrahepatic islet number required for insulin independence of obtaining, with a threshold dose of 9,000 IEQ/kg body weight of the recipient and a maximum sequence number of 3 infusions. The patient will receive after transplantation immunosuppressive therapy with Thymoglobulin for induction, Prograf and Cellcept, both of which are given throughout the duration of the study
  Interventions: Procedure: Allogeneic transplantation of intrahepatic islet

INTERVENTIONS:
Procedure: Allogeneic transplantation of intrahepatic islet

SUMMARY:
It is a multicentre, sequential, phase II clinical trial, aiming at evaluating the allogeneic islet transplantation for the treatment of type 1 diabetes.

19 patients with type 1 diabetes will be included and ideally distributed evenly: patients with unstable diabetes without renal insufficiency (AI group for "islet alone" by the international customary determination) and patients with a functioning kidney transplant (IAK group for "islet after kidney"). The main endpoint will be defined by the restoration of normal glycemic control without insulin at 6 months after graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes
* 18 <Age <55 years
* Plasma C-peptide <0.2 ng/ml basal and stimulated glucagon
* Evolution of diabetes for more than 5 years
* Regular patient follow-up (> or equal to 2 visits per year from the same diabetologist)
* Patient who received the information and have given their consent in writing
* Absence of HIV, hepatitis B and hepatitis C, HTLV-1-2
* ABO compatibility with the donor
* Cross match negative
* Anti-HLA antibodies (class I and / or class II) detected by lymphocytotoxicity <20%
* PCR negative for the BK virus in the blood (so as not to amplify the BK virus replication with the ATG).
* Accepting patients effective contraception during the study period

For patients in group IA

* Glomerular filtration rate estimated by the MDRD> 50 ml/min/1.73m2
* No perception of hypoglycaemia (less than 0.54 mg/dl glucose) at least one value documented in the two years preceding and/or
* Occurrence of at least one severe hypoglycemic episode (with a third required) and unexplained in the two years before and/or at least two episodes of ketoacidosis per year
* Average HbA1c> 8.5% over two years, despite intensified treatment (basal pattern, bolus)

  • For patients in the IAK
* functional renal graft for at least 1 year
* glomerular filtration rate> 50 ml/min/1.73 m2
* proteinuria <0.5 g/day
* Absence of acute rejection in renal previous 6 months

Exclusion Criteria:

* BMI > 28
* Need insulin > 1 U/kg per day
* Pregnancy, lactation
* Intention of childbearing for the two sexes
* Psychiatric Disorders
* Inability to communicate or cooperate with the investigator
* Lack of therapeutic compliance, including HbA1C > 12%
* Chronic liver disease
* Progressive heart disease myocardial infarction within 6 months prior to inclusion, unbalanced CHD)
* Proliferative retinopathy unstabilized
* History of cancer, whatever the date, except for basal or squamous cell skin cancers over 1 year.
* Systemic infection
* Chronic high risk of requiring corticosteroids
* Need for long-term corticosteroid, outside that specified in renal transplantation, the patients will be weaned before transplantation
* Anticoagulant vitamin K or antiplatelet treatments
* Disorders of hemostasis TP <60 % TCA > 1.5 times the control
* Anti-HLA antibodies ( class I and/or class II ) detected by lymphocytotoxicity > 20%
* Platelets < 100 giga/L and/or neutrophils <1.5 giga/L
* Chronic intoxication by alcohol, tobacco, or other substance (abstinence > 6 months required)
* Active infection by hepatitis B, hepatitis C and HIV, HTLV-1-HTLV2
* Ascites

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
restoration of normal glycemic control without insulin | 6 months after graft
  the restoration of normal glycemic control without insulin therapy will be evaluated by measuring
  - A fasting glucose (> 8 hours) less than 1.25 g/L and a 2 hours glucose after oral intake of 75g of glucose, less than 2 g/L in a patient without insulin for at least 15 consecutive days during the the first 6 months from day 0.

SECONDARY OUTCOMES:
Restoration of normal glycemic control without insulin for a year | 1 year
Obtaining an improvement in glycemic control | within 2 years after inclusion
  HbA1c <6.5%, with lower insulin doses by 30%
Obtaining a remission of diabetes | within 2 years after inclusion
  The remission of diabetes is defined by the normality of blood glucose or insulin without lHbA1c.
  The normality of blood glucose is defined below 1.20 g/L and postprandial fasting glycemia less than 1.60 g/L in the book self-monitoring (including 6/7 blood glucoses during the previous 3 days evaluation visit).
  Normal HbA1c is defined as less than 6.5%.
Improved metabolic profile determined by the OGTT and hyperglycemic clamp | within 2 years after inclusion
Decreased glycemic variability | within 2 years after inclusion
  defined on blood glucose and / or glucose holter
Reduction of oxidative stress assessed by the urinary excretion of 24 hours of 8-iso-PGF2 rates. | within 2 years after inclusion
Decrease in the frequency, severity or poor perception of hypoglycaemia defined Hypo score | within the 2 years after inclusion
quality of life | within 2 years after inclusion
  defined by questionnaires DQOL and SF-36
term graft survival | within 2 years of inclusion
  defined by the rate of C-peptide
beta-cell function | 2 years
  based on beta-score
potential of each infusion of islets | within 2 years after inclusion
  number of IEQ/kg of recipient required to reduce the daily insulin dose of 1 unit
degenerative complications of diabetes | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, Île-de-France Region, France